CLINICAL TRIAL: NCT05842564
Title: Autophagic Activity Characterization in Pediatric Crohn's Disease
Brief Title: Autophagy in Paediatric Crohn's Disease
Acronym: P-IBDphagy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL21_1020
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease; Pediatric Crohns Disease
Keywords: Crohn's Disease; Autophagy; Polymorphism
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crohn's Disease Group (Experimental): Patients followed for a Crohn's Disease in consultation or in day hospital aged between 6 and 18 years old.
  Interventions: Other: Blood samples; Other: Biopsies
- Control Group (Other): Patients followed for functional abdominal disorders
  Interventions: Other: Blood samples; Other: Biopsies

INTERVENTIONS:
Other: Blood samples — Blood sample of maximum 20ml (5 tubes of EDTA of 4ml or 5 tubes of EDTA of 2ml and a tube for the conservation of genomic DNA)
Other: Biopsies — 5 biopsies (one for each segment of the intestine explored: ileum, right colon, transverse colon left colon and sigmoid) will be taken during the ileocolonoscopy

SUMMARY:
Crohn's disease is a multifactorial complex disease resulting in a between microbiota and immune system. Indeed, GWAS (Genome-Wide Association Studies) association study pinpointed polymorphisms as genes susceptibility on more than 200 loci. Among them genes coding for proteins involved in autophagy machinery (i.e: ATG16L1, IRGM et NDP52). Autophagy is a ubiquitous intracellular mechanism mandatory for protein and microorganism recycling.

So far, the role of autophagy in gut inflammation and intestinal homeostasis in Crohn's disease patients is partially understand. Then, investigators plan to evaluate, on native cells, the autophagic flux in pediatric patients suffering of a Crohn's disease compare to controls.

ELIGIBILITY:
Inclusion Criteria:

For Crohn's Disease group :

* Age between 6 and 17 inclusive
* Patients with a weight > 25 kg at the time of inclusion
* Patients with Crohn's disease requiring ileocolonoscopy (diagnosis or follow-up)
* Mild to severe Crohn's disease consistent with PCDAI disease activity score
* Patients on nutritional therapy (Modulen/Modulife), corticosteroids, salicylic derivatives, immunosuppressants, biotherapies (anti-TNF, vedolizumab and ustekinumab) or without treatment
* Consent form signed by the patient or the holder(s) of parental authority.
* Affiliation to a social security scheme or beneficiaries of a similar scheme.

For Control group:

* Between 6 and 17 years old included
* Presenting a weight > 25 kg at the time of inclusion
* Without a diagnosis of Crohn's disease
* Requiring evaluation by ileoendoscopy
* Consent form signed by the patient or the holder(s) of parental authority.
* Affiliation to a social security scheme or beneficiaries of a similar scheme.

Exclusion Criteria:

* Refusal to participate in the protocol
* Intercurrent infection
* Ongoing antibiotic treatment
* Patient involved in another interventional study protocol including an exclusion period still in progress at pre-inclusion
* Pregnant, parturient or breastfeeding women (on questioning)
* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Persons admitted to a health or social establishment for purposes other than research

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quantification of autophagic flux by western blot. | 1 day (during hospitalization for ileocolonoscopy)
  LC3II/LC3I will be measured by western blot after booking the autophagic flux at different time point.

SECONDARY OUTCOMES:
Incidence of autophagic polymorphisms in pediatric Crohn's disease population | 1 day (during hospitalization for ileocolonoscopy)
  DNA sequencing of polymorphisms reported in the literature as gene mutations susceptibility for Crohn's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Hépatologie, Gastroentérologie et Nutrition pédiatrique, Hôpital Femme Mère Enfant, HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No